CLINICAL TRIAL: NCT02884401
Title: Radiographic Peri-implant Alveolar Bone Changes in Post-menopausal Osteoporotic Women
Brief Title: Peri-implant Bone Changes in Post-menopausal Osteoporotic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010890
Record Dates: First submitted 2016-06-07; First posted 2016-08-31 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- osteoporotic women with a missing tooth (Other): Post-menopausal osteoporotic women with a missing tooth and willing to replace it with a dental implant
  Interventions: Device: Dental implant placement (Straumann® Bone Level Tapered, BLT, Roxolid® SLActive®)

INTERVENTIONS:
Device: Dental implant placement (Straumann® Bone Level Tapered, BLT, Roxolid® SLActive®) — A tapered bone level implant (Straumann® BLT Roxolid® SLActive®, Basel, Switzerland) will be placed according to the manufactures guidelines trying to achieve primary stability in the correct prosthetic position

SUMMARY:
This is a prospective case series study aiming to evaluate the effect of post-menopausal osteoporosis on the jaw bone around dental implants with a modified titanium surface. The study consists of 8 visits that will be performed within a minimum period of 15 months. Participants will be recruited from the Rheumatology Department and Radiology Department at Barts Health National Health Service (NHS) Trust.

Participants will include 20 post-menopausal osteoporotic women with a requirement of a tooth to be replaced. The main objective of this study is to radiographically compare alveolar (jaw) bone changes in width and height after the placement of a dental implant with a hydrophilic (SLActive) surface and 12 months after loading (placement of the crown) it in post-menopausal osteoporotic women.

DETAILED DESCRIPTION:
This is a prospective case series study aiming to radiographically assess the changes in alveolar bone width and height after the placement of a SLActive implant (implant with a modified surface that should stimulate bone formation) and 12 months after loading it in post-menopausal osteoporotic women. The null hypothesis is: in post-menopausal osteoporotic women there are no significant changes in the peri-implant alveolar bone after the placement of a SLActive implant and 12 months after loading it in terms of width and height assessed by the use of CBCT images. The aim is to include 20 post-menopausal osteoporotic women with a requirement of a tooth to be replaced. However, considering a potential drop-out rate of 10%, the investigators have planned to increase the recruitment for this trial to 22 postmenopausal women. They will be recruited from the Rheumatology Department and Radiology Department at Barts Health NHS Trust, amongst those patients attending for a consultation with the osteoporosis specialist or for taking a Dual-energy X-ray absorptiometry (DXA) scan. Before starting the visit, post-menopausal women meeting the inclusion criteria will be asked by a study examiner if they agree to be quickly screened for the presence of an intercalate edentulous area (edentulous area in between the teeth)and if they may be interested in taking part into the study. If they agree, a quick dental examination will be performed by a study examiner (a qualified dentist) after the visit. The patients who would qualify for enrolment will receive information on the study, the patient information sheet and consent form, together with a letter to give to their General Dental Practitioner (GDP) in order to be referred to the Centre for Oral Clinical Research. The patients that do not qualify for enrolment will receive a report of the oral screening in case they require dental treatments.

Once the referral letter arrives at the Centre for Oral Clinical Research, Barts Health, the patient will be contacted to answer any further question and to book an appointment to attend the enrolment visit, should they wish.

The study consists of 8 visits that will be performed over a minimum period of 15 months at the Centre for Oral Clinical Research at the School of Dentistry of Queen Mary University of London (QMUL):

1. Enrollment visit:

   * Signing of informed consent;
   * Recording of any concomitant medication;
   * Confirmation of participant eligibility pertaining to the presence of an intercalate single edentulous area fulfilling the inclusion criteria (wisdom teeth and second molars excluded)
   * Basic Periodontal Examination (BPE) recording;
   * Clinical measurement of the periodontal parameter in the teeth adjacent to the area where the implant will be placed (Probing pocket Depth, PPD; Recession, REC; Plaque Index, PI; Bleeding on Probing, BOP)
   * Exit participant if not eligible, arrangement for full-mouth debridement treatment outside the study protocol (if needed) and refer to GDP for other dental problems (such as caries and endodontic infections).

   If the patient agrees, a letter will be sent to the General Practitioner (GP) to inform about the participation in the study.
2. Full-mouth debridement(within 90 days from enrolment):

   * Recording of any Adverse Event (AE) or concomitant medication;
   * Oral hygiene instructions and supra and sub gingival debridement of all teeth (as necessary) using ultrasonic and hand instruments as indicated. Local anaesthesia may be used as required to ensure pain control for the participant.

   In case a participant requires further periodontal treatment, this will be arranged outside the study protocol. No implant will be placed until a condition of periodontal health (no pockets ≥5 mm) will be reached.

   • In order to plan the implant placement and according to the clinician's judgment and the complexity of the case, either a Cone Bean Computed Tomography (CBCT) scan or a peri-apical intra-oral x-ray, limited at the area of the implant placement, will be taken.
3. Implant placement (within 120 days from visit 2):

   * Recording of any AE or concomitant medication;
   * Implant placement. If required, simultaneous horizontal guided regeneration (GBR) of the alveolar bone with a collagen membrane (Collprotect®, Botiss®, Zossen, Germany) and a bovine osteoconductive graft (Cerabone, Botiss®, Zossen, Germany) will be performed;
   * Recording of maximum torque at placement;
   * Healing cap screwed for semi-submerged healing;
   * Resonance frequency analysis;
   * Standardized CBCT scan limited to the implant area No sinus lift cases will be taken into consideration.
4. Suture removal (7 days + 3 days from Visit 3):

   * Recording of any AE or concomitant medication;
   * Clinical evaluation of soft tissue healing (visual inspection of the surgical site and report of any complication);
   * Suture removal;
   * Resonance frequency analysis;
   * Standardized CBCT scan limited to the implant area (if not performed on the day of implant placement).
5. Implant impression (6 weeks ± 7 days from Visit 3):

   * Recording of any AE or concomitant medication;
   * Implant impression;
   * Resonance frequency analysis. In case horizontal GBR is performed simultaneously to implant placement, the implant impression will be performed 11 weeks (+7 days) after implant placement.
6. Implant loading (8 weeks ± 7 days from Visit 3):

   * Recording of any AE or concomitant medication;
   * Clinical measurement of the periodontal parameter in the teeth adjacent to the implant (PPD, REC, PI, BOP);
   * Implant loading and occlusion control;
   * Resonance frequency analysis;
   * Peri-apical X-ray In case GBR is performed simultaneously to implant placement, the implant impression will be performed 12 weeks (+7 days) after implant placement.
7. 6-months follow-up (6 months ± 14 days from Visit 6):

   * Recording of any AE or concomitant medication;
   * Clinical measurement of the periodontal parameter in the teeth adjacent to the implant (PPD, REC, PI, BOP) and on the implant
   * Polish and oral hygiene instructions;
   * Resonance frequency analysis;
8. 12-months follow-up (12 months ± 14 days from Visit 6):

   * Recording of any AE or concomitant medication;
   * Clinical measurement of the periodontal parameter in the teeth adjacent to the implant (PPD, REC, PI, BOP) and on the implant;
   * Polish and oral hygiene instructions;
   * Resonance frequency analysis;
   * CBCT scan and evaluation of implant survival and success. Photos of the teeth/implant may be taken to facilitate case documentation. The photos will be strictly limited to the implant/teeth area so that subjects will not be identifiable.

At study completion, a letter will be sent to the patient's GDP to inform about the treatments provided and highlight any need for further treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must present a diagnosis of osteoporosis based on DXA measurement of the bone mineral density at the femur neck and/or total hip and/or lumbar spine (T value 2.5 SD or more below the young female adult mean) within the past 24 months.
* Not in treatment with anti-resorptive agents (like bisphosphonates and denosumab) for more than 4 consecutive years, in order to reduce the risk of medication-related osteonecrosis of the jaws (Lo et al., 2010).
* ≥ 50 years old.
* In self-reported menopause, defined as the permanent cessation of ovulation, for at least one year (Soules et al., 2001).
* Edentulous area involving a maximum of two teeth (wisdom teeth and second molars are excluded) and presenting at least one neighbouring tooth (e.g. gap in the area of a second premolar and first molar, with first premolar in place).
* Residual alveolar width ≥ 4 mm (Milinkovic and Cordaro, 2014), residual alveolar height >8 mm, enough inter-arch space for a crown (at least 5 mm) and a minimum distance of 7 mm from the adjacent teeth (Shah and Lum, 2008). The width and height will be confirmed after x-ray examination in Visit 2.
* Possibility to restore a functional occlusion with a minimum of four occlusal units (i.e. pairs of occluding posterior teeth).
* Willingness to replace the missing tooth/teeth with dental implants
* Registration with a GDP

Exclusion Criteria:

* On chronic treatment (i.e., two weeks or more) with any medication severely affecting oral status (e.g. participants with gingival hypertrophy caused by anti-epileptics, calcium antagonists, cyclosporine and other immunosuppressive) or bone metabolism (e.g. anticoagulant medications, long-standing steroid medications -i.e. equal or more 2.5mg of prednisolone a day taken for >3 months -, anticonvulsants, immunosuppressants).
* Affected by systemic diseases recognized to severely affect bone metabolism (e.g. Cushing's syndrome, Addison's disease, diabetes mellitus type 1, leukaemia, pernicious anaemia, malabsorption syndromes, chronic liver disease, rheumatoid arthritis).
* Knowingly affected by HIV or Hepatitis.
* History of local radiation therapy in the last five years.
* Affected by limited mental capacity or language skills such that study information cannot be understood, informed consent cannot be obtained, or simple instructions cannot be followed.
* Presenting an acute endodontic/periodontal lesion in the neighboring areas to the implant site.
* Completely edentulous
* With evident severe atrophy of the alveolar ridge that could preclude an implant placement (e.g. sharp knife edge ridge)
* Severe bruxism or clenching habits
* Smokers of > 5 cigarettes a day.
* A daily alcohol intake >2 units/day.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality which may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial.
* Patients unable or not willing to return for follow-ups.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in peri-implant horizontal and vertical alveolar bone | After implant placement (+10 days) and 12 months after implant loading (± 14 days)
  The peri-implant alveolar bone changes in height and width (in mm) will be assessed with the use of a CBCT scan after the implant placement (+10 days) and 12 months post loading (± 14 days). A single calibrated examiner will take all the measurements 3 times and the average value will be recorded. All measurements will be calculated with a 0.1 mm precision level.

SECONDARY OUTCOMES:
changes in implant stability measured with resonance frequency analysis | at implant placement, suture removal (7 days + 3 days after implant placement), implant impression (6 weeks ± 7 days after implant placement), implant loading (8 weeks ± 7 days after implant placement), at 6 months- (± 14 days) and 12 months- follow ups.
  Resonance frequency analysis will be used to evaluate implant stability. Implant stability quotient (ISQ) will be recorded after implant placement, suture removal (7 days + 3 days after implant placement), implant impression (6 weeks ± 7 days after implant placement), implant loading (8 weeks ± 7 days after implant placement), at 6 months- (± 14 days) and 12 months- follow ups.
Implant success | 12 months after loading (± 14 days)
  Buser et al (1990) criteria will be used to evaluate implant success 12 months after loading (± 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, Prof, Principal Investigator — Queen Mary University of London
Locations (1):
- Centre for Oral Clinical Research, Institute of Dentistry, Barts Health, QMUL, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buser D, Broggini N, Wieland M, Schenk RK, Denzer AJ, Cochran DL, Hoffmann B, Lussi A, Steinemann SG. Enhanced bone apposition to a chemically modified SLA titanium surface. J Dent Res. 2004 Jul;83(7):529-33. doi: 10.1177/154405910408300704. PMID 15218041
- [Background] Calciolari E, Donos N, Park JC, Petrie A, Mardas N. A systematic review on the correlation between skeletal and jawbone mineral density in osteoporotic subjects. Clin Oral Implants Res. 2016 Apr;27(4):433-42. doi: 10.1111/clr.12597. Epub 2015 Apr 12. PMID 25864584
- [Background] Dao TT, Anderson JD, Zarb GA. Is osteoporosis a risk factor for osseointegration of dental implants? Int J Oral Maxillofac Implants. 1993;8(2):137-44. PMID 8359868
- [Background] Donos N, Hamlet S, Lang NP, Salvi GE, Huynh-Ba G, Bosshardt DD, Ivanovski S. Gene expression profile of osseointegration of a hydrophilic compared with a hydrophobic microrough implant surface. Clin Oral Implants Res. 2011 Apr;22(4):365-72. doi: 10.1111/j.1600-0501.2010.02113.x. PMID 21561478
- [Background] Lang NP, Salvi GE, Huynh-Ba G, Ivanovski S, Donos N, Bosshardt DD. Early osseointegration to hydrophilic and hydrophobic implant surfaces in humans. Clin Oral Implants Res. 2011 Apr;22(4):349-56. doi: 10.1111/j.1600-0501.2011.02172.x. PMID 21561476
- [Background] Mardas N, Schwarz F, Petrie A, Hakimi AR, Donos N. The effect of SLActive surface in guided bone formation in osteoporotic-like conditions. Clin Oral Implants Res. 2011 Apr;22(4):406-15. doi: 10.1111/j.1600-0501.2010.02094.x. Epub 2011 Feb 8. PMID 21303420
- [Derived] Elena C, Nikos M, Iro P, Sara T, Nikolaos D. Radiographic Peri-Implant Bone Changes in Osteoporotic Women Treated With a Ti-Zr, Bone Level Tapered Implant With a Hydrophilic Surface: A 12-Month Prospective Case-Series. Clin Oral Implants Res. 2025 Oct;36(10):1234-1247. doi: 10.1111/clr.14469. Epub 2025 Jul 8. PMID 40625220